NCT : 1690/KEPK/XII/2019

: The Effect of Combination Therapy Using Li-ESWT and PDE-5 Inhibitor Compared to PDE-5 Inhibitor Alone in Patients With Erectile Dysfunction Title

Date : June 14, 2020

| KOMORBID | Dislipidemia, Stroke | HT, Smoking | DM, HT | DM, HT, Dislipidemia | | Gastritis | Ma | HNP, Vertigo | Stone, LOH, Alcoholism, Smoking | DM, HT, Dislipidemia, LOH,<br>Smoking | DM, HT, Heart Disease, CKD<br>on HD, Hiperuricemia, LOH,<br>Smoking, Dislipidemia | DM, Stroke, Merokok | Dislipidemia, LOH | Hernia | Stroke, Dislipidemia, Smoking | HT, STD | DM, Hiperuricemia | Heart disease, Smoking | Hernia | DM, HT, Heart disease,<br>Meningitis | TB, Hepatitis, HT, Heart<br>disease, Smoking, Alcoholism | DM, HT, Heart disease, HNP,<br>BPH | Dislipidemia, LOH | | | HT, Dislipidemia, Smoking |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| BMI<br>(kg/m2) | 25.1 | 22.0 | 33.5 | 27.1 | 23.3 | 26.4 | 23.3 | 23.3 | 31.2 | 27.2 | 32.2 | 29.0 | 31.5 | 22.2 | 30.5 | 32.5 | 27.9 | 24.6 | 18.2 | 26.5 | 18.2 | 23.5 | 29.0 | 29.3 | 26.1 | 30.1 |
| WAIST<br>CIRCUMFERRENCE<br>(cm) | 84 | 68 | 111 | 92 | 68 | 06 | 91 | 92 | 102 | 97 | 113 | 102 | 102 | 75 | 102 | 112 | 66 | 92 | 75 | 101 | 73.5 | 66 | 95 | 100 | 87 | 103 |
| MARRIAGE<br>DURATION<br>(Years) | 12 | 22 | 17 | 29 | 7 | 23 | 19 | 24 | 32 | 25 | 32 | 24 | 21 | 14 | 22 | 18 | 29 | 19 | 11 | 27 | 20 | 25 | 19 | 56 | 30 | 35 |
| AGE OF<br>SPOUSE | 37 | 20 | 48 | 54 | 40 | 41 | 46 | 42 | 52 | 38 | 52 | 40 | 45 | 36 | 48 | 48 | 51 | 46 | 30 | 50 | 37 | 09 | 45 | 53 | 49 | 51 |
| AGE | 40 | 54 | 47 | 54 | 43 | 45 | 48 | 44 | 53 | 48 | 52 | 49 | 49 | 44 | 54 | 47 | 20 | 43 | 46 | 51 | 43 | 53 | 47 | 55 | 53 | 51 |
| ED<br>DURATIO<br>N (Years) | 5.00 | 1.50 | 1.00 | 0.25 | 0.25 | 9.00 | 1.50 | 0.67 | 2.00 | 0.67 | 0.33 | 1.50 | 6.50 | 2.00 | 0.50 | 5.00 | 0.67 | 0.50 | 0.50 | 5.00 | 1.00 | 10.00 | 2.00 | 2.00 | 2.00 | 00.9 |
| ED<br>SEVERITY<br>(Years) | plim | mild | plim | mild | mild-<br>moderate | mild | mild-<br>moderate | mild-<br>moderate | mild | mild-<br>moderate | mild-<br>moderate | mild | moderate | moderate | mild | mild | moderate | mild | moderate | moderate | moderate | moderate | mild | mild | mild-<br>moderate | mild-<br>moderate |
| IIEF5 PRE | 17 | 17 | 17 | 17 | 14 | 20 | 16 | 15 | 19 | 16 | 12 | 16 | 10 | 6 | 19 | 18 | 10 | 21 | 10 | 10 | 10 | 11 | 20 | 17 | 16 | 12 |
| EHS PRE | 2 | 2 | 3 | 2 | 2 | 3 | 2 | 2 | 2 | 2 | ю | 2 | 2 | 1 | 2 | 3 | 1 | 3 | 1 | 1 | 2 | 2 | 3 | 2 | 2 | 2 |
| INITIAL | ELB | RUD | ANZ | BIL | YUD | EDI | ЕДН | SAM | MBA | ALI | SAP | TRI | SAT | MAM | GOD | НОТ | KHO | ROC | MAD | FIR | EDD | ЕКО | BNA | EDO | RAT | PAR |
| GROUP | 1 | 1 | 2 | 1 | Н | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 2 | 2 | 1 | 2 | 2 | 2 | ₽ | 2 |
| <u>Q</u> | 1 | 2 | 3 | 4 | 5 | 9 | 7 | 8 | 6 | 11 | 12 | 13 | 14 | 16 | 17 | 20 | 21 | 22 | 23 | 24 | 25 | 56 | 27 | 28 | 29 | 30 |

Notes : Kelompok 1 = control group (single therapy) Kelompok 2 = test group (combination therapy)

| :HS | | | | | | | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Delta EHS | 1 | 1 | 1 | 1 | 1 | 1 | 7 | 7 | 7 | 1 | 2 | 1 | 2 | 0 | 2 | 1 | 7 | 0 | 7 | 2 | 1 | 1 | 1 | 7 | 7 | 2 |
| Posttest EHS | 3 | 3 | 4 | 3 | 3 | 4 | 4 | 4 | 4 | 3 | 4 | 3 | 4 | 1 | 4 | 4 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 4 | 4 | 4 |
| Pretest EHS | 2 | 2 | 3 | 2 | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 3 | 1 | 3 | 1 | 1 | 2 | 2 | 3 | 2 | 2 | 2 |
| Delta IIEF5 | 3 | 4 | 2 | 2 | 3 | 2 | 6 | 7 | 9 | 2 | 12 | 2 | 15 | 0 | 4 | 7 | 11 | 1 | 14 | 4 | 6 | ∞ | 3 | 4 | 6 | 13 |
| Posttest<br>IIEF5 | 20 | 21 | 22 | 19 | 17 | 25 | 25 | 22 | 25 | 23 | 25 | 21 | 25 | 6 | 23 | 25 | 21 | 22 | 24 | 14 | 19 | 19 | 23 | 21 | 25 | 25 |
| Pretest IIEF5 | 17 | 17 | 17 | 17 | 14 | 20 | 16 | 15 | 19 | 16 | 13 | 16 | 10 | 6 | 19 | 18 | 10 | 21 | 10 | 10 | 10 | 11 | 20 | 17 | 16 | 12 |
| Delta Pre-<br>Post VEGF | 2.44 | -14.65 | 16.92 | -21.30 | -3.43 | 43.13 | 0.36 | 36.96 | 14.05 | 52.84 | 37.38 | 21.78 | 30.18 | 7.78 | 8.23 | -9.88 | 10.26 | -16.43 | 5.72 | 10.17 | 67.14 | 92.73 | 35.82 | 10.97 | 37.67 | 8.23 |
| Posttest<br>VEGF | 100.11 | 137.96 | 81.39 | 61.72 | 53.49 | 139.18 | 24.32 | 80.17 | 100.33 | 93.99 | 67.56 | 77.33 | 70.64 | 79.77 | 45.95 | 14.08 | 82.21 | 70.64 | 26.75 | 102.15 | 173.77 | 159.94 | 134.71 | 69.95 | 52.12 | 69.27 |
| Pretest VEGF | 97.67 | 152.61 | 64.47 | 83.02 | 56.92 | 96.05 | 23.96 | 43.21 | 86.28 | 41.15 | 30.18 | 55.55 | 40.46 | 71.99 | 37.72 | 23.96 | 71.95 | 87.07 | 21.03 | 91.98 | 106.63 | 67.21 | 68.86 | 58.98 | 14.45 | 61.04 |
| Delta Pre-<br>Post PSV | 06.0 | 0.20 | 2.30 | 09.9 | 1.75 | 3.00 | 4.50 | -0.25 | 2.05 | 3.85 | 3.15 | 0.35 | 3.55 | 0.75 | -0.20 | 1.00 | 2.65 | -0.15 | 4.80 | 1.70 | 0.40 | 1.90 | 2.45 | 1.25 | 1.15 | 2.15 |
| Pretest PSV Posttest PSV | 11.10 | 14.20 | 13.00 | 20.80 | 11.35 | 14.00 | 16.15 | 9.00 | 14.95 | 17.95 | 13.95 | 8.85 | 11.75 | 8.70 | 15.30 | 16.50 | 7.85 | 14.50 | 12.70 | 12.40 | 8.95 | 13.00 | 14.90 | 14.25 | 14.05 | 14.40 |
| Pretest PSV | 10.20 | 14.00 | 10.70 | 14.20 | 9.60 | 11.00 | 11.65 | 9.25 | 12.90 | 14.10 | 10.80 | 8.50 | 8.20 | 7.95 | 15.50 | 15.50 | 5.20 | 14.65 | 7.90 | 10.70 | 8.55 | 11.10 | 12.45 | 13.00 | 12.90 | 12.25 |
| GROUP | 1 | н | 2 | 1 | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 2 | 2 | 1 | 2 | 2 | 2 | 1 | 2 |
| INITIAL | ELB | RUD | ANZ | BIL | AND | EDI | HQ3 | SAM | MDA | ALI | SAP | TRI | SAT | MAM | GOD | HOT | КНО | ROC | MAD | FIR | EDD | EKO | BNA | EDO | RAT | PAR |
| Q | 1 | 2 | 3 | 4 | 5 | 9 | 7 | 8 | 6 | 11 | 12 | 13 | 14 | 16 | 17 | 20 | 21 | 22 | 23 | 24 | 25 | 26 | 27 | 28 | 29 | 30 |

Notes : Group 1 : control group (single therapy) Group 2 : test group (combination therapy)

**Table 1.** Subjects characteristics

| Tuble 1: Subjects chara | | Control | Experimental | | |
|---|---|---|---|---|---|
| Characteristics | | Group | Group | Total | p |
| | | n=12 | n=14 | n=26 | |
| Mean Age | | 47.8 yo | 49.2 yo | 48.6 yo | 0,419 |
| Mean Spouses' age | | 44.7 yo | 45.9 yo | 45.3 yo | 0,620 |
| Mean Duration of ED | | | | 2.6 | |
| (years) | | 1.7 years | 3.4 years | years | 0.147 |
| Mean of waist | | | | | |
| circumference | | | | | |
| (cm) | | 91.4 | 97.9 | 94.9 | 0.118 |
| Mean BMI | | | | | |
| $(kg/m^2)$ | | 25.7 | 27.5 | 26.7 | 0.277 |
| Comorbidities | Diabetes Mellitus | 25% | 42.9% | 34.6% | |
| | Hypertension | 33.3% | 42.9% | 38.5% | |
| | Cardiac problems | 16.7% | 21.4% | 19.2% | |
| | Dyslipidemia | 25% | 50% | 38.5% | |
| | Hypogonadism | 0% | 35.7% | 19.2% | |
| | History of smoking | 41.7% | 28.6% | 34.6% | |
| | History of alcoholism | 8.3% | 7.1% | 7.7% | |
| | Other | 50% | 57.1% | 53.8% | |
| ED Severities | Mild | 58.3% | 35.7% | 46.2% | |
| | Mild-Moderate | 16,7% | 35.7% | 26.9% | |
| | Moderate | 25% | 28.6% | 26.9% | |
| Median of EHS | | 2 | 2 | 2 | 0.573 |
| | | (1-3) | (1-3) | (1-3) | 0.573 |
| Median of IIEF-5 | | 16.5 | 15.5 | 16 | 0.716 |
| | | (9-21) | (10-20) | (9-21) | 0.710 |

Note: n = number of samples, ED = erectile dysfunction, BMI = body mass index, EHS = erection hardness score, IIEF = International index of erectal function
Comparison of IIEF-5, EHS, and mean duration of ED were done using Mann-Whitney test, as for other parameters, Independent T-test were used.

**Table 2.** Comparison of IIEF-5 scores

| _ | | Pre-test – Post-test | | |
|---|---|---|---|---|
| Subject | Pre-test | Post-test | Delta | Comparison<br>p |
| Control Group (n=12) | 16.5<br>(9-21) | 21<br>(9-25) | 4<br>(0-12) | 0.004* |
| Experimental Group (n=14) | 15.5<br>(10-20) | 23.5<br>(14-25) | 7<br>(3-15) | 0.001* |
| Total<br>(n=26) | 16<br>(9-21) | 22<br>(9-25) | 5.5<br>(0-15) | |

Note: IIEF=International index of erectile function, n=number of sample, \*= sign of significance (p < 0.05)

Comparison of pre- and post-test IIEF-5 parameter was done using Wilcoxon's test

Table 3. Comparison of EHS scores

| | | Pre-test – Post-test | | |
|---|---|---|---|---|
| Subject | Pre-test | Post-test | Delta | Comparison<br>p |
| Control Group<br>(n=12) | 2<br>(1-3) | 3<br>(1-4) | 1<br>(0-2) | 0.004* |
| Experimental Group (n=14) | 2<br>(1-3) | 4 (3-4) | 2<br>(1-2) | 0.001* |
| Total | 2 | 3.5 | 1 | |
| (n=26) | (1-3) | (1-4) | (0-2) | |

Note: EHS = Erection hardness score, n = number of sample, \* = sign of significance (p < 0.05)

Comparison of pre- and post-test EHS parameter was done using Wilcoxon's test

**Table 4.** Comparison of VEGF values

| | | VEGF Level | | Pre-test – Post-test |
|---------------|----------|------------|-------|----------------------|
| Subject _ | | Comparison | | |
| | Pre-test | Post-test | Delta | p |
| Control Crown | 59.92 | 66.24 | 6.32 | |
| Control Group | ± | ± | ± | 0.408 |
| (n=12) | 41.91 | 49.42 | 25.43 | |
| Experimental | 57.95 | 84.65 | 26.69 | |
| Group | ± | ± | 土 | 0.001* |
| (n=14) | 25.92 | 40.71 | 24.23 | |
| Total | 58.86 | 76.15 | 17.29 | |
| Total | ± | ± | 土 | |
| (n=26) | 33.52 | 44.99 | 26.40 | |

Note: VEGF = Vascular Endothelial Growth Factor, n = number of sample, \* = sign of significance (p < 0.05) Comparison of pre- and post-test VEGF parameter was done using Paired T-test.

**Table 5.** Comparison of PSV values

| | | PSV | | Pre-test - Post-test |
|---------------|----------|------------|-------|----------------------|
| Subject | | Comparison | | |
| | Pre-test | Post-test | Delta | p |
| Control Group | 11.40 | 12.68 | 1.28 | 0.044 |
| Control Group | ± | ± | ± | 0.04* |
| (n=12) | 3.47 | 3.90 | 1.86 | |
| Experimental | 11.14 | 13.74 | 2.60 | 0.001# |
| Group | ± | ± | ± | 0.001* |
| (n=14) | 1.79 | 2.10 | 1.34 | |
| Total | 11.26 | 13.25 | 1.99 | |
| | 土 | 土 | ± | |
| (n=26) | 2.64 | 3.04 | 1.70 | |

Note: PSV = Peak Systolic Velocity, n = number of sample, \* = sign of significance (p < 0.05)

Comparison of pre- and post-test PSV parameter was done using Paired T-test.

**Table 6.** Comparison of all parameters between groups

| | rameter | Control Group | Experimental Group | p |
|--------|-----------|-------------------|--------------------|--------|
| | Pre-test | 16.5 (9-21) | 15.5 (10-20) | 0.716 |
| IIEF-5 | Post-test | 21 (9-25) | 23.5 (14-25) | 0.047* |
| | Delta | 4 (0-11) | 7 (3-15) | 0.047* |
| | Pre-test | 2 (1-3) | 2 (1-3) | 0.573 |
| EHS | Post-test | 3 (1-4) | 4 (3-4) | 0.018* |
| | Delta | 1 (0-2) | 2(1-2) | 0.032* |
| | Pre-test | $59.92 \pm 41.91$ | $57.95 \pm 25.92$ | 0.885 |
| VEGF | Post-test | $66.24 \pm 49.42$ | $84.65 \pm 40.71$ | 0.308 |
| | Delta | $6.32 \pm 25.43$ | $26.69 \pm 24.23$ | 0.023* |
| | Pre-test | $11.40 \pm 3.47$ | $11.14 \pm 1.79$ | 0.813 |
| PSV | Post-test | $12.68 \pm 3.90$ | $13.74 \pm 2.10$ | 0.385 |
| | Delta | $1.28 \pm 1.86$ | $2.60 \pm 1.34$ | 0.009* |

Note: IIEF = International index of erectile function, EHS = Erection hardness score, PSV = Peak Systolic Velocity, VEGF = Vascular Endothelial Growth Factor, \* = statistically significant (p < 0.05)

Comparison between groups for pre-test and post-test VEGF parameters were done using Independent T-test, as for the others parameters, the statistics methods used was Mann-Whitney test